CLINICAL TRIAL: NCT04873726
Title: Effects of Magnetic Tape on Autonomic Nervous System in Patients With Low Back Pain
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Logistics and infrastructure problems
Sponsor: Francisco Selva (Other)
Responsible Party: Sponsor-Investigator, Francisco Selva, Principal Investigator, Clínica Dr. Francisco Selva
Organization: Clínica Dr. Francisco Selva (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 5
Record Dates: First submitted 2021-04-26; First posted 2021-05-05 (Actual); Last update posted 2022-09-14 (Actual); Status verified 2022-09

CONDITIONS: Low Back Pain
Keywords: low back pain; pupil; Magnetic tape®; pinch; Vorteq® system; autonomic nervous system; pain; algometer
MeSH Terms: conditions — Low Back Pain; Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (9):
- Pre: pain AP (No Intervention): Pain assessment in the spinous processes of the spine with algometer anteroposterior pressure
- Pre: pain Pinch test (No Intervention): perceived pain over the paravertebral skin at each level of the spine using Pinch test
- Pre: pupil diameter (No Intervention): the pupil responses were measured with the fully automated Vorteq® system (Micromedical Technologies, Inc) to record the pupil reaction.
- Post Exp: pain AP (Experimental): Pain assessment in the spinous processes of the spine with algometer anteroposterior pressure
  Interventions: Device: Magnetic Tape® aplication
- Post Exp: pain Pinch test (Experimental): perceived pain over the paravertebral skin at each level of the spine using Pinch test
  Interventions: Device: Magnetic Tape® aplication
- Post Exp: pupil diameter (Experimental): the pupil responses were measured with the fully automated Vorteq® system (Micromedical Technologies, Inc) to record the pupil reaction.
  Interventions: Device: Magnetic Tape® aplication
- Post Pla: pain AP (Placebo Comparator): Pain assessment in the spinous processes of the spine with algometer anteroposterior pressure
  Interventions: Device: Kinesiology Tape
- Post Pla: pain Pinch test (Placebo Comparator): perceived pain over the paravertebral skin at each level of the spine using Pinch test
  Interventions: Device: Kinesiology Tape
- Post Pla: pupil diameter (Placebo Comparator): the pupil responses were measured with the fully automated Vorteq® system (Micromedical Technologies, Inc) to record the pupil reaction.
  Interventions: Device: Kinesiology Tape

INTERVENTIONS:
Device: Magnetic Tape® aplication — Magnetic tape® is applied without creating any tension on the lumbar paravertebral skin to assess changes in pupil size
  Arms: Post Exp: pain AP; Post Exp: pain Pinch test; Post Exp: pupil diameter
Device: Kinesiology Tape — Kinesiology tape is applied without creating any tension on the lumbar paravertebral skin to assess changes in pupil size
  Arms: Post Pla: pain AP; Post Pla: pain Pinch test; Post Pla: pupil diameter

SUMMARY:
The tape will be applied on the lumbar area bilateralemten to the spine without creating any tension.

Possible variation in the autonomic nervous system is assessed in the reaction of the pupils. A kinesiology tape was used as a placebo tape and the magnetic tape was used in a randomized experimental way.

DETAILED DESCRIPTION:
A triple-blind cross-sectional observational study is designed where subjects with low back pain will be selected and blinded to recieve the Magnetic Tape® (tape with magnetic effects of less than 2 Gauss) or placebo Tape. Likewise, the evaluator who puts the Magnetic Tape® does not know what material he is using, as it is supplied by another researcher. The statistician will also be blinded.

The recommendations of the "Reporting of Observational Studies in Epidemiology" (STROBE) will be followed. All participants will receive a participant information sheet and sign informed consent. Patients aged 18 to 65 years with low back pain will be recruited from different private clinics in the city of Valencia, Spain.

The hypothesis is that when Magnetic Tape® comes into contact with electromagnetic fields such as those generated by living beings, due to the movement of electrical charges (ions), as defined by Ampere's Law, the domains of the tape are oriented or aligned in parallel with the external magnetic field creating a magnetic flux with a north pole and a south pole. This generated field in turn produces a magnetic induction proportional to the variation of the magnetic flux, as defined by the Faraday Law.

This electric potential produces a redistribution of the electric charge (ions) generating a magnetic field due to the orientation of the tape domains, then exerting a force on the moving charges within the electrolyte.

Physiological, Lorentz's Law, regulating Magnetic Tape® aberrant electromagnetic fields.

After signing the informed consent and data protection, the groups with low back pain will be formed that will receive the application of both Magnetic Tape® and the intervention of a placebo tape. To avoid that the order of the intervention influences the results of the study, the subjects will be randomized into two different groups, Group A and Group B. Group A will receive Magnetic tape® and Group B will do the opposite. The next day the other tape will be applied.

The patient will be placed in the prone position and the spinous processes of T11 and L5 will be identified by marking them with a pen. Once L4 is located at the level of the iliac crests, the therapist will palpate the following spinous processes and will count down to the level of T11 and L5, and then mark it.

Later two strips of tape will be placed on the lumbar paravertebral skin. To measure ANS activity during this study the vortex from Micromedical will be used to capture the pupil diameter. Each participant will wear the goggles throughout the measurement phase and will be in a prone position (with the eyes in complete darkness). After the goggles are placed properly the subjects will remain in a quiet room for three minutes to accommodate to the room environment before the pupil measurement. After this, a 60 second pupil recording will be taken. This measurement will serve as the participant's baseline measurement. After the tape placement the pupil will immediately measured again for a duration of 60 seconds. After a 30 second break period in which the subject is able to blink and close the eyes a second 60 second measure of the pupil will be taken. These steps will be repeated so there will be a total of 4 post measure 60 second pupil measurements (post measure 1, 30 sec break, post measure 2, 30 sec break, post measure 3, 30 sec break, post measure 4). Regardless of what tape is used that will be the measurement sequence.

After signing the subject informed consent and data protection groups will be formed. There will be two groups. The first group will consist of spinal pain patients. This group will receive both a Magnetic Tape®, and the placebo tape intervention. The second group without back pain will be age matched to the spine group and will receive the Magnetic Tape®. The spine pain patients are given the two interventions on two different days and wills serve as their own control. To prevent the order of the intervention to influence the study results the subjects will be randomized into two different groups, Spine A and Spine B. Spine A will receive the Magnetic Tape® on their first visit and receive a kinesiology tape on their next visit. Spine B will do the opposite. The control group will only receive the intervention tape.

After this, the subject will be placed on a treatment table in the prone position. In this position, a physical therapist will provide posterior to anterior pressure applied at the spinous process and the segmental skin pinch test and it will be documented whether this pressure would cause any pain. If any pain is reported, the subject will be asked to rate this pain on a Numerical Pain Rating Scale (NPRS). The pressure was carried out from S3 to C2.

Neither application has to be painful.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with low back pain.
* Subjects aged 18-65 years.

Exclusion Criteria:

* Tape allergies
* Adhesive allergies
* Pregnant
* People with pacemakers
* People who have any contraindication of electromagnetic fields
* Peoplewith neurological diseases
* Taking any medication that may interact with magnetic fields.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-07-22 (Estimated); Primary Completion 2022-12-22 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Pressure | Changes from pressure on spinous processes, first assessment before placing the tapes and inmediatly after placing experimental tape and placebo tape
  pressure in each spinous process
Pupil reaction | Changes from pupil diameter, first assessment before placing the tapes and inmediatly after placing experimental tape and placebo tape
  the pupil responses were measured with the fully automated Vorteq® system (Micromedical Technologies, Inc)
Pinch test | Changes from paravertebral pinch test, first assessment before placing the tapes and inmediatly after placing experimental tape and placebo tape
  press the paravertebral skin at each level of the spine with the first three fingers

CONTACTS AND LOCATIONS:
Locations (1):
- Clinica Francisco Selva, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No